CLINICAL TRIAL: NCT01526200
Title: Factors Influencing the Impact of Contrast-Enhanced Intraoperative Ultrasound During Liver Surgery for Colorectal Cancer Liver Metastases
Brief Title: Contrast-Enhanced Intraoperative Ultrasound During Liver Surgery for Colorectal Cancer Liver Metastases
Acronym: CEIOUSCLM
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Professor of Surgery, MD, PhD, University of Milan
Other Study IDs: CEIOUSCLM
Record Dates: First submitted 2012-01-27; First posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-01

CONDITIONS: Colon Cancer Liver Metastasis
Keywords: CLM
MeSH Terms: interventions — contrast agent BR1; Sonazoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CEIOUS: One hundred and twenty-seven consecutive patients -77 males and 50 females, mean age of patients was 61 years (median 65 years; range 29-85 years)- underwent liver resection using intraoperative ultrasound and contrast-enhanced intraoperative ultrasound.
  Interventions: Procedure: Contrast-enhanced intraoperative ultrasound

INTERVENTIONS:
Procedure: Contrast-enhanced intraoperative ultrasound — After entering the abdominal cavity, liver mobilization is achieved by dissecting the round and falciform ligaments. IOUS is carried out with a standard 3-6 MHz convex probe, and a 7.5-10 MHz micro convex probe. Staging was completed by CE-IOUS using the standard 3-6 MHz convex probe and the dedicated 1.88-3.76 MHz harmonic frequency probe. In all patients, 2.4 mL of sulphur-hexafluoride microbubbles (SonoVue®, Bracco, Milan, Italy) are injected through a peripheral vein by the anesthesiologist.
  Other Names: Sonovue, Sonazoid, CEIOUS

SUMMARY:
Contrast-enhanced intraoperative ultrasound (CE-IOUS) during surgery for colorectal liver metastases (CLM) has become a part of clinical practice. However, if it should be selectively or routinely applied remains unclear. This study is carried out to clarify which are the criteria for a selective use of CE-IOUS if any.

DETAILED DESCRIPTION:
Contrast-enhanced intraoperative ultrasound (CE-IOUS) during surgery for colorectal liver metastases (CLM) is entered in clinical practice. However, its impact seems to decrease with the improvement of preoperative imaging. Therefore, if CE-IOUS should be selectively or routinely applied remains unclear: a profile of patients who may benefit of CE-IOUS application has to be disclosed. The aim of this study is to define reliable criteria for a selective use of CE-IOUS during surgery for CLM. IOUS is performed using 3-6 MHz convex probe, and a 7.5-10 MHz micro convex probe. Staging is completed by CE-IOUS using the standard 3-6 MHz convex probe and the dedicated 1.88-3.76 MHz harmonic frequency probe. In all patients, 2.4 mL of sulphur-hexafluoride microbubbles (SonoVue®, Bracco, Milan, Italy) are injected through a peripheral vein by the anesthesiologist. Ultrasound guidance is used to drive the dissection plane as previously described. Reference standards are histology and imaging at 6 months after surgery. Univariate and multivariate analyses are performed. Statistical significance is set at P=0.05.

ELIGIBILITY:
Inclusion Criteria:

* consecutively enrolled patients with CLM who underwent surgery and during this procedure received IOUS and CE-IOUS.
* each patient had at least 6 months of postoperative follow-up.

Exclusion Criteria:

* patients who after IOUS and CE-IOUS had explorative laparotomy only were excluded from the analysis since there was no histological confirmation of the tumor and most of them were lost to surgical follow-up

Ages: 29 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutively enrolled patients with CLM who underwent surgery and during this procedure received IOUS and CE-IOUS.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2007-10; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
new colorectal liver metastases detected at contrast-enhanced intraoperative ultrasonography | October 2007 - March 2011 (up to 4 years)

SECONDARY OUTCOMES:
new colorectal liver metastases detected at intraoperative ultrasonography | October 2007 - March 2011 (up to 4 years)
new colorectal liver metastases detected during 6-month postoperative follow-up | October 2007 - December 2011 (up to 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Principal Investigator — University of Milano
Locations (1):
- Istituto Clinico Humanitas IRCS, Rozzano, Milan, Italy